CLINICAL TRIAL: NCT06165302
Title: EPC Trial: Exercise in Prostate Cancer
Brief Title: Exercise in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Physical Medicine & Rehabilitation Educ Research Foundation, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J23147; IRB00410196 (Other: JHM IRB)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer
Keywords: Exercise Intervention
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Participants will be prescribed an exercise program after completing assessments at baseline. Participants will adhere to the prescribed exercise intervention for 12 weeks and log activity in a physical activity diary. Participants will return to clinic on Week 5 and Week 9 for assessments and adjustment to their exercise prescription as needed.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — 12 weeks of prescribed exercise intervention.

SUMMARY:
The goal of this clinical trial is to learn how exercise intervention affects circulating tumor cells (CTC) in men with advanced prostate cancer. The primary objective is to determine if an exercise intervention decreases CTCs in men with advanced prostate cancer. Participants will have baseline screening assessments, followed by 12 weeks of exercise intervention, and then follow-up assessments 12 weeks after the end of the exercise intervention.

DETAILED DESCRIPTION:
This is a pilot single arm prospective study of personalized exercise training in men with metastatic castration resistant prostate cancer who are being treated with or without oral anti-androgens. The primary objective is to determine if combination of resistance and aerobic exercises lowers CTCs in men with mCRPC. Researchers will assess the rate of conversion from CTC positive to CTC negative in participants at the end of the 12 week exercise intervention. The study will enroll 20 participants onto the trial with the goal of at least 10 participants having blood drawn at both baseline and 12 weeks and completed at least 75% of the prescribed exercise sessions. Participants will undergo follow-up assessments at the end of the 12 week exercise intervention and the study team will monitor participant records for 365 days after the study completion for vital status.

ELIGIBILITY:
Inclusion Criteria:

1. Men with metastatic prostate adenocarcinoma
2. Currently taking androgen deprivation therapy alone or with an oral androgen axis inhibitor (abiraterone, enzalutamide, darolutamide, or apalutamide are permitted) and have been on treatment for at least 3 months
3. Elevated (PSA > 1ng/mL) or rising PSA (any numerical increase based on at least 2 PSA readings at least 2 weeks apart)
4. Any number of prior therapies (prior chemo, radium-223, etc.) is allowed
5. CTC + according to standard clinical grade laboratory test by androgen receptor isoform splice variant 7 (AR-V7) testing at Hopkins.
6. If a bone protective agent is to be started, it should be started at least 2 weeks prior to the onset of exercise intervention.
7. Eastern Cooperative Oncology Group (ECOG) performance status <=1
8. Clearance by cardiologist if under the current care of a cardiologist (seen in the past 1 year)
9. Age <=80 years

Exclusion Criteria:

1. Small cell carcinoma of the prostate
2. Unable to participate or monitor exercise compliance due to conditions such as impaired cognition
3. Moderate to severe bone pain that limits any activities of daily living, including use of narcotics for prostate cancer related pain
4. Clinical progression requiring a change in systemic therapy or the addition of palliative radiation for symptom control
5. Bone metastases in spine or long bones which, in the eye of the treating physician require referral to radiation oncology or surgery for management due to risk of fracture
6. Significant cardiovascular disease or concurrent illness that would make exercise intervention for 12 weeks unsafe. If there is significant cardiovascular disease and the participant is under the care of a cardiologist (seen within the past 1 year), approval of the cardiologist to participate is required.
7. Major surgery within the past 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with negative CTC count | Baseline, 12 weeks
  Number of participants with negative CTC count at 12 weeks compared to the baseline

SECONDARY OUTCOMES:
Number of participants with change in cell free DNA levels | Baseline, 12 weeks
  Number of participants with change in cell free DNA levels from baseline to 12 weeks
Number of participants with change in Cell free RNA levels | Baseline, 12 weeks
  Number of participants with change in cell free RNA levels from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Marshall, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No